CLINICAL TRIAL: NCT01087151
Title: A Phase II, Multicenter, Randomized, Controlled, Open-label Study of the Safety, Efficacy and Pharmacokinetics of ABT-263 in Combination With Dose-intensive Rituximab, or Dose-intensive Rituximab Alone, in Previously Untreated Patients With B-Cell, Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study of ABT-263 in Combination With Dose-Intensive Rituximab, or Dose-Intensive Rituximab Alone, in Previously Untreated Patients With B-Cell, Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT4710n; 2009-012152-24 (EudraCT Number); GP00763 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-03-11; First posted 2010-03-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Rituxan; Apoptosis; BCl-2
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — navitoclax; Rituximab

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: rituximab
- B (Experimental)
  Interventions: Drug: ABT-263; Drug: rituximab
- C (Experimental)
  Interventions: Drug: ABT-263; Drug: rituximab

INTERVENTIONS:
Drug: ABT-263 — Oral repeating dose
  Arms: B; C
Drug: rituximab — Intravenous repeating dose

SUMMARY:
This Phase II, randomized, open-label, international, multicenter trial is designed to evaluate the safety and efficacy of rituximab monotherapy when given according to a dose intense regimen and to assess the safety, efficacy, and pharmacokinetics of ABT-263 when combined with dose-intense rituximab in previously untreated patients with B-cell CLL.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, CD20-positive B-cell CLL
* ECOG performance status of 0 or 1
* Life expectancy > 6 months
* Willingness and capability to be accessible for follow-up until study termination or death
* For patients of reproductive potential (both males and females), use of a reliable means of contraception

Exclusion Criteria:

* Prolymphocytic leukemia
* Richter's transformation to an aggressive B-cell malignancy (e.g., DLBCL)
* Prior radiotherapy to a lesion(s) that will be used to assess response unless that lesion(s) shows clear evidence of progression at baseline
* Patients with a history of other malignancies within 2 years prior to study entry except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin carcinoma, low-grade, localized prostate cancer treated surgically with curative intent or one that carries a good prognosis, in situ ductal carcinoma of the breast treated with lumpectomy alone with curative intent
* Prior treatment with rituximab, ABT-263 or other pro-apoptotic agents
* Current or recent (within the 28 days prior to initiation of study treatment) participation in another experimental drug study
* Major surgical procedure (excluding lymph node biopsy) or significant traumatic injury within 28 days prior to treatment onset or anticipation of the need for major surgery during the course of the study
* Active infection requiring parenteral antibiotics or antiviral or antifungal agents at the onset of study treatment
* Receipt of primary or booster vaccination with live-virus vaccines for up to 6 months prior to initiation of study treatment
* Patients receiving therapeutic anticoagulation with heparin or warfarin or patients receiving any drugs or herbal supplements that are known to inhibit platelet function (including low-dose aspirin) within 7 days of the first dose of ABT-263. Note: Patients receiving low-dose anticoagulation for the purpose of maintaining central venous catheter patency are eligible.
* Patients who have an inherited or acquired bleeding diathesis, including (but not limited to) hemophilia or immune or thrombotic thrombocytopenic purpura, or who have had an underlying condition that predisposes to abnormal bleeding (e.g., peptic ulcer disease) within 1 year prior to the first dose of ABT-263
* Patients with a history of refractoriness to platelet transfusions
* Clinically significant cardiovascular disease
* Known human immunodeficiency virus (HIV) infection, seropositivity for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody or RNA
* Pregnancy or breastfeeding
* Concurrent (or within 7 days prior to the first dose of study treatment) systemic corticosteroid therapy except some low-dose corticosteroid therapies
* History of other disease, metabolic dysfunction, physical or laboratory finding(s) giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, might affect interpretation of the results of the study or render the patient at high risk from treatment complications
* History of anaphylaxis, allergic reaction, or hypersensitivity to sulfites (sodium metabisulphite is included in study drug formulation)
* Any contraindication to alcohol ingestion (study drug formulation includes approximately 15% ethanol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From randomization to the first occurrence of progression, relapse, or death on study (approximately 40 months from First Patient In [FPI])

SECONDARY OUTCOMES:
Overall response rate (ORR) | Approximately 40 months from FPI
Duration of response | Approximately 40 months from FPI
Complete response (CR) rate | Approximately 40 months from FPI
Progression-free survival as assessed by a blinded, independent review | From randomization to the first occurrence of progression, relapse, or death on study (approximately 40 months from FPI)
ORR as assessed by a blinded, independent review | Approximately 40 months from FPI
Duration of response as assessed by a blinded, independent review | Approximately 40 months from FPI
CR rate as assessed by a blinded, independent review | Approximately 40 months from FPI
Overall survival (OS) | From randomization until death due to any cause (approximately 4 years after Last Patient In)

CONTACTS AND LOCATIONS:
Overall Officials: William Ho, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (92):
- United States (41):
  - Alhambra, California
  - Antioch, California
  - Berkeley, California
  - Burbank, California
  - Duarte, California
  - Dublin, California
  - La Jolla, California
  - Los Angeles, California
  - Northridge, California
  - Pleasant Hill, California
  - San Leandro, California
  - San Luis Obispo, California
  - Santa Monica, California
  - Fort Collins, Colorado
  - Norwalk, Connecticut
  - Bay Pines, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Decatur, Illinois
  - Harvey, Illinois
  - Tinley Park, Illinois
  - Shreverport, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Randallstown, Maryland
  - Lansing, Michigan
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Reno, Nevada
  - Cherry Hill, New Jersey
  - Farmington, New Mexico
  - Oneida, New York
  - Oswego, New York
  - Syracuse, New York
  - Middletown, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Corpus Christi, Texas
  - Lubbock, Texas
  - Everett, Washington
- Australia (9):
  - Randwick, New South Wales
  - Greenslopes, Queensland
  - Adelaide, South Australia
  - Kurralta Park, South Australia
  - Coburg, VIC, Victoria
  - Fitzroy, Victoria
  - Frankston, Victoria
  - Parkville, Victoria
  - Fremantle, Western Australia
- Brazil (7):
  - Cachoeiro de Itapemirim, Espírito Santo
  - Belo Horizonte, Minas Gerais
  - Rio de Janeiro, Rio de Janeiro
  - Caxias do Sul, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São Paulo, São Paulo
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- France (2):
  - Lille
  - Pierre-Bénite
- Israel (4):
  - Afula
  - Petah Tikva
  - Ramat Gan
  - Rehovot
- Italy (6):
  - Modena, Emilia-Romagna
  - Genoa, Liguria
  - Cremona, Lombardy
  - Milan, Lombardy
  - Rozzano, Lombardy
  - Turin, Piedmont
- Poland (3):
  - Chorzów
  - Gdansk
  - Warsaw
- San Juan, Puerto Rico
- Russia (5):
  - Kazan'
  - Moscow
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
- Ukraine (9):
  - Cherkassy
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Khmelnitskyy
  - Kyiv
  - Lviv
  - Poltava
  - Zhytomyr
- United Kingdom (2):
  - Leicester
  - London